CLINICAL TRIAL: NCT07386821
Title: The Effect of Laughie Exercise on Pain Anxiety and Pain Level in Second-Degree Burn Patients: A Randomised Controlled Trial
Brief Title: Effect of Laughie on Pain Anxiety and Pain Level in Second-Degree Burn Patients
Acronym: LA-PAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Burcu Duluklu, Asst. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TABED 2-25-1864
Record Dates: First submitted 2026-01-25; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Burn; Second Degree Burns
Keywords: burn; laughie; pain; pain anxiety
MeSH Terms: conditions — Burns; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Laughie
  Interventions: Other: Laughie
- Control Group (No Intervention): Control:
  Second-degree burn patients. For patients presenting for their second dressing change, standard dressing change prosedures will be applied. The study procedure will include the following steps: (1) collection of descriptive characteristics; (2) assessment of pain severity and pain anxiety levels 5-10 minutes before the dressing change; (3) application of the dressing; (4) reassessment of pain severity and pain anxiety levels five minutes after the procedure.

INTERVENTIONS:
Other: Laughie — One alternative and complementary medicine approach that has gained attention is the Laughie technique, also known as guided laughter exercise. Laughie enables individuals to laugh in a controlled manner using their own voice, targeting the physiological and psychological benefits of laughter.
  In this study, Laughie involves recording a one-minute video of the patient's natural laughter. Before the dressing change, patients watch this video and accompany their laughter to support autonomic nervous system stabilization.
  For patients presenting for their second dressing change, the study procedure will include the following steps: (1) collection of descriptive characteristics; (2) assessment of pain severity and pain anxiety levels 5-10 minutes before the dressing change; (3) administration of the Laughie exercise five minutes before the dressing change; (4) application of the dressing; and (5) reassessment of pain severity and pain anxiety levels five minutes after the procedure.
  Arms: Intervention Group

SUMMARY:
Burn injuries are traumatic conditions that seriously affect individuals' quality of life, both physically and psychologically. Second-degree burns, in particular, affect the superficial and/or deep layers of the dermis, causing intense pain and extensive tissue damage. Pain in burn patients is not only physical; it combines with emotional stress, fear, and uncertainty to increase anxiety levels.

This study is a parallel group-randomised controlled trial designed to evaluate the effects of the Laughie exercise, administered prior to dressing changes in individuals diagnosed with second-degree burns, on post-dressing pain anxiety levels and pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over
* Having a second degree burn
* Arriving for the second dressing change on the unit
* To agree to participate in the research

Exclusion Criteria:

* In multiple burns, a burn degree other than the second degree on any part of the body
* A maximum of 96 hours have elapsed since the burn injury
* To have come to the dressing in repetitions other than the second dressing
* Inability to tolerate the Laughie exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
1. Burn Specific Pain Anxiety | Change from baseline scores at the end of 15 minutes.
  The Burn Specific Pain Anxiety Scale (BSPAS) consists of nine items. The scale was designed to assess pain-related anxiety in patients with burn injuries. The Turkish version includes eight items, each rated on a two-ended visual analog scale ranging from 0 to 10, with anchor points defined as "none at all" (0) and "in the worst possible way" (10). Total scores are calculated by summing the item scores, yielding a possible range from 0 to 80. Higher total scores reflect greater levels of pain-related anxiety experienced by patients during painful hospital procedures. The internal consistency of the Turkish version was excellent, with a Cronbach's α coefficient of 0.95.

SECONDARY OUTCOMES:
The Visual Analog Scale (VAS) | Change from baseline scores at the end of 15 minutes.
  The Visual Analog Scale (VAS) is a widely used, simple, and reliable tool for assessing subjective experiences such as pain intensity. It typically consists of a 10-cm horizontal or vertical line anchored by two endpoints representing extreme states, ranging from "no pain" to "worst imaginable pain." Patients are asked to indicate the point that best reflects their current level of pain, providing a quantitative measure of pain severity that is easy to administer and sensitive to change.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Duluklu, PhD, Asst. Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No